CLINICAL TRIAL: NCT04341571
Title: Effect of the Administration of Probiotics Versus Metformin on Glycemic Control, Insulin Sensitivity and Insulin Secretion in Patients With Prediabetes.
Brief Title: Effect of Probiotics Versus Metformin on Glycemic Control, Insulin Sensitivity and Insulin Secretion in Prediabetes.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Karina Griselda Pérez Rubio, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Probiotics-Prediabetes
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: PreDiabetes; Impaired Glucose Tolerance; Hyperglycemia; Resistance, Insulin
Keywords: Probiotics; Prediabetes; Hyperglycemia; Impaired Fasting Glucose; Glucose intolerance; Metformin
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Hyperglycemia; Insulin Resistance | interventions — Probiotics; Metformin

STUDY DESIGN:
Intervention Model Description: Double-blind, controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: Randomized double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): 15 patients to receive homologated intervention capsule (probiotics lactobacillus acidophilus y bifidobacterium lactis 400 mg) 1 time at day before breakfast along 13 weeks and receive 1 homologated placebo capsule (calcinated magnesia 500 mg) 1 time at day before dinner along 13 weeks.
  Interventions: Dietary Supplement: Probiotics
- Metformin (Experimental): 15 patients to receive homologated intervention capsule (metformin 750 mg) twice at day before breakfast and dinner for 13 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotics capsules (lactobacillus acidophilus y bifidobacterium lactis) 400 mg 1 time at day before breakfast and one placebo capsule before dinner during 13 weeks. Homologated to the other intervention.
  Arms: Probiotics
Drug: Metformin — Metformin capsules, 750 mg, two pere day before breakfast and dinner during 13 weeks.
  Homologated to the other intervention.
  Arms: Metformin

SUMMARY:
Pre diabetes (PD) is a term that refers to alterations in blood glucose levels, including impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or both, and increase in glycated hemoglobin (HbA1c), all this factors involving a higher risk to develop type 2 diabetes mellitus (T2DM).

The efficacy of pharmacotherapy in the prevention of diabetes in adults with pre diabetes has been demonstrated, the first line of pharmacology treatment is metformin, on the other hand, probiotics administration has been reported to be one of the most widely used approaches to modulate the gut microbiota and subsequently prevent or delay the incidence of T2DM.

Probiotics are live microorganisms which when administered in adequate amounts confer a health benefit on the host. Has been demonstrated the hypoglycemic effects of the probiotics in different clinical trials in type 2 diabetes mellitus and pre diabetes, but no yet compared with metformin, for this reason comparing it´s activity against metformin in pre diabetes would provide impact information on a new alternative treatment compared with the standard pharmacological treatment.

The aim of the study is evaluate the effect of administration of probiotic versus metformin on glycemic control, insulin secretion and insulin sensitivity in patients with pre diabetes.

DETAILED DESCRIPTION:
A randomized, double-blind controlled clinical trial in 30 patients between 31 to 60 years of age with a diagnosis of prediabetes (IFG 100 a 125 mg/dL, IGT 140 a 199 mg/dL, HbA1c 5.7 a 6.4%) in accordance with the American Diabetes Association without treatment.

Patients with one or more of the following criteria will be excluded: History of liver, kidney or heart disease; systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg, HbA1c ≥6.5%, triglycerides ≥ 400 mg/dL, total cholesterol ≥240 mg/dL; pregnancy or lactation; consumption of medications or supplements with effects on glucose levels.

They will be assigned randomly two groups of 15 patients; one of the groups will receive 750 mg of metformin twice at day (before breakfast and dinner) for 13 weeks.

The other group will receive 400 mg of probiotics 1 time at day (before breakfast) and placebo pill (before dinner) for 13 weeks.

They will be measured fasting blood glucose, postprandial glucose levels and glycosylated hemoglobin, and will be calculated area under curve of glucose an insulin, total insulin secretion (Insolinogenic index), first-phase of insulin secretion (Strumvoll index) and insulin sensitivity (Matsuda index).

This protocol It´s already approved by the local ethics committee and written informed consent it´s going to be obtained from all volunteers.

Statistical analysis will be presented through measures of central tendency and dispersion, average and deviation standard for quantitative variables; frequencies and percentage for qualitative variable. Will be used Wilcoxon range test for identification of differences between baseline and final evaluation of each intervention group, Mann-Whitney U Test and Wilcoxon Test for the within-groups differences. It will be considered satitistical significance p >0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 31 and 60 years
* Diagnosis of prediabetes according ADA criteria (fasting blood glucose levels between 100-125 mg/dL, postprandial blood glucose levels after an oral glucose tolerance test with 75 g of oral glucose between 140-199 mg/dL and glycated hemoglobin between 5.7-6.4 %)
* Body Mass Index from 25 to 34.9 kg/m2
* Stable weight at least the previous last 3 months (weight variation less than 10%)
* Acceptance and signing of informed consent

Exclusion Criteria:

* History of kidney, liver or heart disease
* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Physical impossibility for taking pills
* Hypersensibility to ingredients of intervention
* Consumption of medications or supplements with effects on glucose levels
* Systolic blood pressure ≥ 140 mmHg
* Diastolic blood pressure ≥ 90 mmHg
* HbA1c ≥6.5%
* Triglycerides ≥ 400 mg/dL
* Total cholesterol ≥ 240 mg/dL

Ages: 31 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose levels | Baseline to week 13 (end of intervention)
  The fasting glucose levels will be evaluated at baseline and week 13 by enzymatic- colorimetric technique to get fasting glucose level
Postpandrial glucose levels | Baseline to week 13 (end of intervention)
  Glucose will be evaluated at baseline and week 13 after a oral glucose tolerance test with enzymatic-colorimetric technique
Glycosylated hemoglobin | Baseline to week 13 (end of intervention)
  Glycosylated hemoglobin will be evaluated at baseline and week 13 by high efficiency liquid chromatography.
Insulin sensitivity | Baseline to week 13 (end of intervention)
  Insulin sensitivity will be calculated at baseline and week 13 with Matsuda index to get insuline sensitivity
Total insulin secretion | Baseline to week 13 (end of intervention)
  Total insulin secretion will be calculated at baseline and week 13 with Insulinogenic index to get total insulin secretion
First phase of insuline secretion | Baseline to week 13 (end of intervention)
  The first phase if insuline secretion will be calculated at baseline and week 13 with Stumvoll index to get first phase of insuline secretion

SECONDARY OUTCOMES:
Body weight | Baseline to week 13 (end of intervention)
  Body weight will be measured at baseline and week 13 with a bioimpedance balance
Body mass index (BMI) | Baseline to week 13 (end of intervention)
  Body mass index will be calculated at baseline and week 13 with the Quetelet index formula
Waist circunference | Baseline to week 13 (end of intervention)
  Waist circunference will be evaluated at baseline and week 13 by World Health Organization technique
Blood pressure | Baseline to week 13 (end of intervention)
  Systolic blood pressure and diastolyc blood pressure will be measured at baseline and week 13 with a digital sphygmomanometer three times in each arm to get an average
Total cholesterol | Baseline to week 13 (end of intervention)
  Total chilesterol level will be evaluated at baseline and week 13 by enzymatic- colorimetric technique to get total cholesterol level
High density lipoprotein (c-HDL) | Baseline to week 13 (end of intervention)
  High density lipoprotein (c-HDL) level will be evaluated at baseline and week 13 by enzymatic- colorimetric technique to get c-HDL level
Low density lipoprotein (c-LDL) | Baseline to week 13 (end of intervention)
  Low density lipoprotein (c-LDL) level will be calculated at baseline and week 13 with Friedewald formula to get c-LDL level
Very low density lipoprotein (VLDL) | Baseline to week 13 (end of intervention)
  Very low density lipoprotein (VLDL) level will be calculated at baseline and week 13 with triglycerides concentration/5 formula to get VLDL level
Fasting blood triglycerides concentration | Baseline to week 13 (end of intervention)
  Fasting blood triglycerides concentration level will be evaluated at baseline and week 13 by enzymatic- colorimetric technique to get triglycerides concentration
Concentration of blood creatinine | Baseline to week 13 (end of intervention)
  Concentration of blood creatinine level will be evaluated at baseline and week 13 by enzymatic-colorimetric technique to get creatinine level
Concentration of blood alanine aminostranferase (ALT) | Baseline to week 13 (end of intervention)
  Concentration of blood alanine aminostranferase level will be evaluated at baseline and week 13 by enzymatic-colorimetric technique to get ALT level
Concentration of blood aspartate aminostranferase (AST) | Baseline to week 13 (end of intervention)
  Concentration of blood aspartate aminostranferase level will be evaluated at baseline and week 13 by enzymatic-colorimetric technique to get AST level
Incidence of treatment-Emergent Adverse Events | Baseline to week 13 (continuous surveiilance)
  Incidence of treatment-Emergent Adverse Events of probiotics+placebo or metformin will be identified by clinical evaluation from baseline week to week 13 with continuous surveiilance

CONTACTS AND LOCATIONS:
Overall Officials: KARINA G PÉREZ-RUBIO, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- INSTITUTO DE TERAPÉUTICA EXPERIMENTAL Y CLÍNICA. Centro Universitario de Ciencias de la Salud, Guadalajara, Jalisco, Mexico